CLINICAL TRIAL: NCT06070220
Title: The Effectiveness of Client-Centered Intervention on Quality of Life and Perceived Occupational Performance and Satisfaction After Total Hip Arthroplasty-A Single Blind Randomized Controlled Study
Brief Title: The Effectiveness of Client-Centered Intervention inTotal Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Berkan Torpil, PhD, Associate Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-53875521
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Hip Osteoarthritis
Keywords: Client-centered; Quality of life; Occupational performance; Hip arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- client-centered intervention group (Experimental)
  Interventions: Behavioral: traditional occupational therapy intervention and client-centered intervention
- control group (Experimental)
  Interventions: Behavioral: Traditional occupational therapy intervention

INTERVENTIONS:
Behavioral: traditional occupational therapy intervention and client-centered intervention — Traditional occupational therapy intervention and client centered intervention were given to the participants.
  CC intervention is a dynamic approach that involves a systematic therapy process, that is, in which the participant and the therapist are active in the treatment process. In the current study, a treatment program was designed over a maximum of 5 occupations in which participants evaluated after THA indicated problems in activities of daily living according to COPM. This systematic and dynamic program consists of 4 phases: (1) client-centered goal setting, (2) negotiating an intervention plan, (3) the actual intervention, (4) an evaluation of the outcome and finally reporting to relevant others.
  Arms: client-centered intervention group
Behavioral: Traditional occupational therapy intervention — The following training procedure, which included exercise, transfer activities and home arrangements, was followed in common in both groups:
  1. st day: After the operation, exercises to strengthen the muscles of the participants (thigh, hip and trunk muscles) were explained verbally and visually. Each exercise consists of 3 sets of 12 repetitions. Exercises were updated in bed, sitting or standing, depending on the participant's functional status, pain and fatigue. Additionally, transfer activities training was provided.
  2. nd day: The exercises taught to the participants on the first day were repeated. Following these exercises, participants were given verbal instructions on gait training, and then gait training began. According to the pain and fatigue status of the participants, gait exercises were continued.
  3. rd day: The work done on the first and second day was repeated. Pre-discharge home arrangements training was provided.
  Arms: control group

SUMMARY:
The current study was conducted to effectiveness of the Client-centered (CC) intervention after Total Hip Arthroplasty (TKA). The current study was planned to examine the impact of the CC intervention on quality of life, perceived occupational performance and satisfaction. The current study was designed according to the CONSORT statement, which provides a standardized method for randomized controlled trial (RCT) design. Approval for the study was granted by the Local Ethics Committee. Written informed consent was obtained from all participants prior to the study.

DETAILED DESCRIPTION:
This study was designed to examine the effectiveness of 6-week CC intervention on quality of life and perceived occupational performance and satisfaction level in individuals aged 65 and over after THA. The study has a randomized controlled structure planned according to the CONSORT Statement. Approval for the study was granted by the Local Ethics Committee. Written informed consent was obtained from all participants prior to the study.

Participants To determine the number of samples, a power analysis, detailed in the statistical analysis section, was performed and it was determined that there should be at least 16 participants for each group. The study evaluated 41 older adults, considering the inclusion and exclusion criteria, as well as predicting participants who would drop out of the study for any reason during the intervention process. These 41 participants who were admitted to a public university's occupational therapy department between July 2022 and July 2023 were screened.

According to the inclusion and exclusion criteria, one participant from each group was excluded from the study because they participated in another rehabilitation program. The remaining 39 participants were randomly assigned to either the CC group or the control group using a computer-generated randomization technique. Initial evaluations were made of the participants, who were divided into 20 participants in the CC group and 19 participants in the control group. Afterwards, during the intervention process, 2 participants from the CC group and 1 from the control group were excluded from the study because they could not participate regularly.

Measurement The demographic characteristics of the participants were recorded, including age, sex, education level, body mass index, smoking/alcohol use, operation region. On the other hand, the following scales were used for all participants, both for use in the inclusion criteria and to measure quality of life and perceived occupational performance and satisfaction.

The scale used in the inclusion criteria:

Mini Mental State Examination In the inclusion criteria, Mini Mental State Examination used to determine cognitive status consists of a maximum of 30 points. 24 points is considered the threshold value, and scores of 24 and above indicate good cognitive skills. Turkish validity and reliability studies of the test have been conducted and the researcher found the Mini Mental State Examination positive and negative predictive values .90 and .95 respectively and kappa score .86.

Scales used in the current study:

Nottingham Health Profile Nottingham Health Profile (NHP) is a 38-item quality of life survey that measures individuals' perceived health problems and the extent to which these health problems affect ADLs.

Canadian Occupational Performance Measure The Canadian Occupational Performance Measure (COPM) was used to identify occupations where participants had problems with ADLs and to determine the perceived occupational performance and satisfaction level in these occupations. In the COPM, which was designed with the semi-structured interview method, firstly, the occupations in which the participants experience problems in the areas of self-care, productivity and free time are determined by giving importance points with a 1-10 Likert type scoring system. Afterwards, a maximum of 5 occupations with the highest importance are determined and the participants give performance and satisfaction scores to these occupations using a 1-10 Likert type scoring method. The performance and satisfaction points given for each occupation are summed and the performance and satisfaction points are divided by the number of occupations received. As a result, participants' perceived occupational performance and satisfaction scores are obtained. The Turkish adaptation performed and test re-test reliability of Turkish version of COPM performance was .988 and satisfaction .986, indicating excellent reliability.

Intervention

This program, which was created before discharge and applied to both groups, was created using the literature. The following training procedure, which included exercise, transfer activities and home arrangements, was followed in common in both groups:

1. st day: After the operation, exercises to strengthen the muscles of the participants (thigh, hip and trunk muscles) were explained verbally and visually. Each exercise consists of 3 sets of 12 repetitions. Exercises were updated in bed, sitting or standing, depending on the participant's functional status, pain and fatigue. Additionally, transfer activities training was provided:

   Transfer Activities Training Considering the needs of the participants, a transfer activities training program was created using the literature. This training program teaches participants how to transfer on wet floors such as toilets and bathrooms, and from one room to another, to beds, chairs, wheelchairs and sofas. Additionally, how to go up and down stairs in a healthy way is explained.
2. nd day: The exercises taught to the participants on the first day were repeated. Following these exercises, participants were given verbal instructions on gait training, and then gait training began. According to the pain and fatigue status of the participants, gait exercises were continued.
3. rd day: The work done on the first and second day was repeated. Pre-discharge home arrangements training was provided:

Home arrangements training Home arrangements training was provided in order to eliminate problems in areas of the house that are difficult to move and may cause injuries such as living room, bathroom, toilet, kitchen, bedroom, corridor, stairs and to perform daily living activities more independently. In this training home injuries and causes of falls, changes that can be made at home, the use of assistive technology, the use of the right adaptive equipment are explained. Home arrangement training to increase mobilization and prevent various injuries such as the use of grab bars, arranging furniture, using adequate lighting (such as using a photocell lamp in the hallway or increasing the light intensity), how to prevent slipping on a wet floor, lifting door sills, moving carpets and cables, using ramps, rearranging seats/chairs/beds to facilitate the transfer process information.

In addition, each participant was given a home visit after discharge and home arrangements were made.

Client-centered intervention The CC intervention was planned to consist of 45-minute sessions 3 days a week for 6 weeks, after the first 4-day rehabilitation procedure given jointly both group.

CC intervention is a dynamic approach that involves a systematic therapy process, that is, in which the participant and the therapist are active in the treatment process. In the current study, a treatment program was designed over a maximum of 5 occupations in which participants evaluated after THA indicated problems in activities of daily living according to COPM. This systematic and dynamic program consists of 4 phases: (1) client-centered goal setting, (2) negotiating an intervention plan, (3) the actual intervention, (4) an evaluation of the outcome and finally reporting to relevant others. A key factor in implementing this intervention program is the problems and priorities prioritized for the participant. The details of the intervention program are described below:

1. st stage: Occupations that cause performance problems in ADLs living should be identified. Realistic and achievable goals for these problems should be designed. In addition, it should be determined how these occupations are affected after THA.
2. nd stage: Brainstorming should be done for possible solutions to the problems experienced in the occupations specified by the participants. Then the pros and cons of the identified solutions should be evaluated.
3. rd stage: Once participants have decided on possible solutions, a plan should be made and action taken. Adaptation of the occupation determined by COPM in terms of time, place, person, how it is done, and the steps of the occupation (in accordance with priority).
4. th stage: The participant should be informed about the progress of the CC intervention and the participant's experiences. If necessary, the intervention should be updated by consensus with the participant.

Statistical Analysis Statistical Package for the Social Sciences software (SPSS v. 28, IBM Corporation, New York, NY, USA) was used for all statistical analyses. The level of significance was set at P < 0.05 and the data are represented as mean±standart deviation. To compare quality of life and occupational performance, an analysis of covariance (ANCOVA) was performed using pre-test values as covariates and post-test values as dependent variables. Before analyzing data, all assumptions of ANCOVA, including normality, homogeneity, homogeneity of regression slopes, and linearity were checked and met. Partial et squared was calculated to assess the effect size, following Cohen's classification where 0.01 represents a small effect, 0.06 stands for a medium effect, and 0.14 indicates a large effect.

ELIGIBILITY:
Inclusion Criteria:

* (1) Being 65 years of age or older,
* (2) Mini Mental State Examination score of ≥ 24,
* (3) having undergone unilateral total hip replacement,
* (4) education level of at least completion of elementary school,
* (5) ability to understand and follow verbal instructions,
* (6) volunteer to participate in the study

Exclusion Criteria:

* (1) revision surgery,
* (2) having any chronic disease that will affect the rehabilitation process,
* (3) auditory and visual problems that may affect rehabilitation implementation and communication,
* (4) postoperative complications (e.g. nerve injury and deep vein thrombosis), and
* (5) attendance of any rehabilitation program (physiotherapy, speech therapy, psychotherapy, etc.) before and during the study period

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure | 40 minutes
  The Canadian Occupational Performance Measure (COPM) was used to identify occupations where participants had problems with ADLs and to determine the perceived occupational performance and satisfaction level in these occupations. In the COPM, which was designed with the semi-structured interview method, firstly, the occupations in which the participants experience problems in the areas of self-care, productivity and free time are determined by giving importance points with a 1-10 Likert type scoring system. The higher the score, the higher the performance and satisfaction level.
Nottingham Health Profile | 10 minutes
  Nottingham Health Profile Nottingham Health Profile (NHP) is a 38-item quality of life survey that measures individuals' perceived health problems and the extent to which these health problems affect ADLs. It consists of 6 sub-dimensions and each sub-dimension consists of 0-100 points (0 points indicate good health status-100 points indicate poor health status): energy (3 items), pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items), and physical activity (8 items). The Turkish version of the NHP was used to evaluate the health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Turkey (Türkiye)